CLINICAL TRIAL: NCT05306821
Title: Effectiveness of Interventions for Hospital Medical Thromboprophylaxis: a Bicentric Swiss Quality-improvement Study
Acronym: TPX-ENHANCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marc Blondon (Other)
Responsible Party: Sponsor-Investigator, Marc Blondon, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-01976
Record Dates: First submitted 2022-02-02; First posted 2022-04-01 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation of an electronic tool for risk stratification and thromboprophylaxis prescription (Experimental)
  Interventions: Other: Comprehensive electronic tool in the electronic medical chart; Other: Educative sessions
- Implementation of educative sessions and pocket cards for thromboprophylaxis (Experimental)
  Interventions: Other: Educative sessions; Other: Pocket card

INTERVENTIONS:
Other: Comprehensive electronic tool in the electronic medical chart — Use of a comprehensive electronic tool in the electronic medical chart to help the stratification of risk of VTE and the subsequent prescription of an adequate thromboprophylaxis
  Arms: Implementation of an electronic tool for risk stratification and thromboprophylaxis prescription
Other: Educative sessions — Educative sessions on thromboprophylaxis
Other: Pocket card — Pocket card (guide for thromboprophylaxis)
  Arms: Implementation of educative sessions and pocket cards for thromboprophylaxis

SUMMARY:
The primary objective is to evaluate and compare the short-term and medicum-term effectiveness of 2 types of interventions in 2 different hospitals to improve the adequacy of hospital thromboprophylaxis among acute medical inpatients.

ELIGIBILITY:
Inclusion Criteria:

* acute medical inpatients hospitalized at the Geneva University Hospitals or the Lugano Regional Hospitals

Exclusion Criteria:

* patients already on therapeutic anticoagulation
* patients with an estimated life expectancy of <3 months
* pregnancy
* patients hospitalized for COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with an adequate thromboprophylaxis | 90 days

SECONDARY OUTCOMES:
Incidence of venous thromboembolism | 90 days
Incidence of major bleeding | 90 days

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Geneva University Hospitals, Geneva
  - Ospedale Regionale di Lugano, Lugano

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marando M, Blondon K, Darbellay Farhoumand P, Nendaz M, Grauser D, Sallet A, Tamburello A, Pons M, Righini M, Gianella P, Blondon M. Contemporary adequacy of thromboprophylaxis in acutely ill medical patients in Switzerland: a bi-centric prospective cohort. Swiss Med Wkly. 2023 Nov 1;153:40117. doi: 10.57187/smw.2023.40117. PMID 37956238